CLINICAL TRIAL: NCT01493375
Title: Surgical Field Bacterial Contamination in Primary Hip and Knee Replacement Surgery
Brief Title: Surgical Field Bacterial Contamination in Primary Total Hip (THA) and Knee (TKA) Arthroplasty
Status: Suspended | Type: Observational
Why Stopped: Study principal investigator left the organization
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); University of Aarhus (Other); Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: N-20100008
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Prosthetic Infections
Keywords: Contamination, hip operation, knee operation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In Denmark, approximately 13,000 operations are carried out every year. Prosthetic infection is a very serious condition and despite extensive prophylactic measures, prosthetic infections appear in 1-2 percent of the operated patients.

It is difficult to diagnose prosthetic infection with the techniques applied so far and incorrect diagnosis might imply unnecessary reoperations as well as unnoticed infections might lead to prolonged pain and invalidity.

The purpose of this study is to examine the value of these three techniques applied as a supplement to the existing technology and on this basis to prepare an algorithm for the examination of joint prosthesis infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been through an alloplastic operation in hip og knee.

Exclusion Criteria:

* Patients with cancer or a bilateral disease
* Former patients who have been through an operation with implants in hip or knee.
* Patients who might be infected in the joint due to operation in hip or knee.
* Lack of informed consent or inability to read/understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Northern Orthopaedic Division, Clinic Frederikshavn.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Contamination of the operation area | 12 months
  We want to examine the existence of contamination before an operation in hip and knee. Furthermore, we want to examine the contamination to achieve better knowledge of the bacterial combination.

SECONDARY OUTCOMES:
Description of the bacterial culture | 12 months
  We want to describe the bacterial culture to achieve better knowledge of the bacterial combination.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Kohler, PhD student, Principal Investigator — Orthopaedic Surgery Research Unit, Aalborg University Hospital; Sten Rasmussen, M.D., Study Director — Northern Orthopaedic Division, Aalborg University Hospital
Locations (1):
- Northern Orthopaedic Division, Clinic Frederikshavn, Frederikshavn, Northern Jutland, Denmark